CLINICAL TRIAL: NCT03807700
Title: A Randomized, Single-blind, Efficacy Study to Evaluate Oral Health and Quality of Life Associated With Use of a Denture Adhesive
Brief Title: To Evaluate Oral Health and Quality of Life Associated With Use of a Denture Adhesive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 209510
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Results first posted 2020-05-01 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Denture Retention
Keywords: Denture, Adhesive, Gum-Health, Lifestyle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental denture adhesive (Experimental): In this arm, participants will apply the experimental adhesive on their dentures once per day when the denture is placed in mouth.
  Interventions: Drug: Experimental Denture Adhesive
- No adhesive (No Intervention): In this arm, participants will not use any denture adhesive.

INTERVENTIONS:
Drug: Experimental Denture Adhesive — In this arm, participants will apply the experimental adhesive on their dentures once per day when the denture is placed in mouth.
  Arms: Experimental denture adhesive

SUMMARY:
The aim of this study is to evaluate the use of a denture adhesive and its ability to demonstrate the improvement in overall gum-health and to improve the oral health related quality of life (OHrQoL) in participants who wear full dentures.

DETAILED DESCRIPTION:
This study will be a single center, controlled, single-blind, randomized, two-treatment, parallel design in healthy participants with a full conventional, acrylic denture in either or both dental arches, with a treatment period of 12 weeks. The study will assess the effectiveness of an experimental denture adhesive in the improvement of denture-bearing tissue irritation related measures, and the participant's oral health related quality of life. Participants will be randomized to one of the 2 treatment groups i.e. experimental denture arm group and control arm group and will undergo an oral soft tissue (OST) examination. Participants with satisfactory dentures, adequate retention and stability and who qualify all the inclusion and exclusion criteria will continue in the study. Participants will complete the Gum Comfort, OHIP-Edent questionnaires and GOHAI questionnaire. The assessments will be made at Baseline, and after 1, 4, 8 and 12 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
2. A participant who is willing and able to comply with scheduled visits, treatment plan, and other study procedures.
3. A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant/relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
4. Pregnant women: must agree to use a highly effective method of contraception throughout the study and for 5 days after the last dose of assigned treatment.
5. Participant has denture prostheses that fulfill all of the following:

   1. A conventional acrylic full denture in either or both of the upper and lower arches. The full denture may be opposed by a partial denture, natural teeth or another full denture.
   2. Dentures are well fitting (Kapur (Olshan Modification) Retention and Stability Index Sum Score ≥ 3 for each denture [maxillary and/or mandibular] with no individual stability or retention scores <1.

   c Denture(s) are well made (according to the well-made assessment).
6. Participant is a habitual wearer of their denture(s) defined as participants who wear their dentures for the majority of their time whilst awake.
7. Participant has worn their full denture(s) for at least a year.
8. Participant has not used any denture adhesive in the last year.
9. Participant currently adopts acceptable denture cleansing habits and routine (a minimum would include daily brushing with a chemical cleaner such as toothpaste or soap, in addition to at least once a week soaking in commercial denture cleansing product). Unacceptable cleaning would include cleaning with water alone or using other non-specialized cleaning methods.

Exclusion Criteria:

1. A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GlaxoSmithKline Consumer Healthcare (GSKCH) employee directly involved in the conduct of the study or a member of their immediate family.
2. A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
3. A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
4. A participant who is a pregnant female.
5. A participant who is a breastfeeding female.
6. A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
7. A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.
8. A participant unwilling or unable to comply with the Lifestyle Considerations:

   1. Participants will not be permitted to have any dental/denture work performed during the time they are in the study, unless discussed and permitted by the examiner. This is to ensure that the denture fit will not be altered during the study.
   2. Participants will not be able to use any denture adhesive product other than that supplied by the investigator.
   3. Participants should continue using their usual denture cleansing methodology throughout the study.
9. A participant who has previously been enrolled in this study.
10. A participant who has had recent (within 30 days) gingival surgery.
11. Taking or have taken a bisphosphonate drug (i.e. Fosamax, Actonel, Boniva).
12. A participant with any clinically significant or relevant oral abnormality (e.g. temporomandibular joint problems) that, in the opinion of the investigator, could affect the Participant's participation in the study.
13. A participant with any condition or medication which, in the opinion of the investigator, is currently causing xerostomia.
14. A participant with recent history (within the last year) of alcohol or other substance abuse.
15. A participant with OST examination findings such as stomatitis, open sores, lesions, or swelling which in the opinion of the investigator, would interfere with the conduct of the study. Mild, chronic conditions commonly expected from the use of dentures in the investigators opinion, are acceptable in this study.
16. A participant who is using any medication that, in the opinion of the investigator, would interfere with the conduct of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-05-04 (Actual); Study Completion 2019-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Mississauga, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a single center in Canada. A total of 119 participants were screened, all of which were enrolled and randomized into the study.
Pre-assignment Details: Participants were allocated to randomized treatment in 2 different arms- experimental adhesive group and no adhesive group.
Groups:
- Experimental Denture Adhesive: In this arm, participants applied denture adhesive in continuous strips to their dentures once per day and then pressed dentures into their mouth and bit firmly to secure the denture hold. Participants recorded their denture cleaning and adhesive application in a study diary for 12 weeks.
- No Adhesive: In this arm participants refrained from using denture adhesive. The participants recorded their denture cleaning occasions in a study diary for 12 weeks.
Period: Overall Study
Arm/Group | Experimental Denture Adhesive | No Adhesive
Started | 60 | 59
Completed | 58 | 58
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Denture Adhesive | No Adhesive | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (9.45) | 67.0 (8.56) | 66.8 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 26 | 61
  Male | 25 | 33 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 58 | 58 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 9 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 7 | 16
  White | 44 | 41 | 85
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Gum Health Analysis by Change From Baseline in Overall Mean Scores of Participant Responses to the Gum Comfort Questionnaire After 12 Weeks
Description: Gum comfort questionnaire was referred to assess the gum health of the denture wearer and to compare the ability of an experimental denture adhesive to provide self-perceived mucosal benefits compared to the use of no adhesive after 12 weeks of product use. It was comprised of 5 questions- Q1: My gums feel comfortable when wearing my denture(s), Q2: I feel my gums are cushioned from the impact of chewing and biting; Q3: My gums do not feel sore at the end of the day; Q4: My gums are not irritated by trapped food particles under my denture(s); Q5: My gums do not feel tired at the end of the day. The participants recorded the response on scale of 0-4: 0-Agree Strongly, 1-Agree Somewhat, 2-Neither Agree or Disagree, 3-Disagree Somewhat, 4- Disagree Strongly). Total score range is 0-20 where lower score indicated better results.
Time Frame: At Baseline and after 12 weeks
Population: Analysis was performed on modified intent-to-treat (mITT) population which included all randomized participants who received at least one dose of study product and had at least one post randomization measure of gum comfort recorded via the questionnaire. Number analyzed included participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 59 | 58
Score on scale
  Baseline | 4.1 (4.22) | 4.5 (3.55)
  Change from baseline after week 12: number analyzed (Participants) | 58 | 58
  Change from baseline after week 12 | -0.6 (3.08) | -0.4 (4.16)
Statistical Analysis 1: Comparison: Experimental Denture Adhesive vs No Adhesive; Test type: Superiority; p = 0.4769, ANCOVA; Analysis was performed using ANCOVA model with study product as a fixed effect and Baseline overall score as a covariate; Mean Difference (Net) = -0.41, 95% CI 2-sided [-1.56 to 0.74], Standard Error of Mean 0.58 — Difference is experimental adhesive minus no adhesive

2. Secondary Outcome: Gum Health Analysis by Change From Baseline in Overall Mean Scores of Participant Responses to the Gum Comfort Questionnaire After 1, 4 and 8 Weeks
Description: Gum comfort questionnaire was referred to assess the gum health of the denture wearer and to compare the ability of an experimental denture adhesive to provide self-perceived mucosal benefits compared to the use of no adhesive after 1, 4 and 8 weeks of product use. It was comprised of 5 questions- Q1: My gums feel comfortable when wearing my denture(s), Q2: I feel my gums are cushioned from the impact of chewing and biting; Q3: My gums do not feel sore at the end of the day; Q4: My gums are not irritated by trapped food particles under my denture(s); Q5: My gums do not feel tired at the end of the day. The participants recorded the response on scale of 0-4: 0-Agree Strongly, 1-Agree Somewhat, 3-Neither Agree or Disagree, 4= Disagree Strongly). Total score range is 0-20 where lower score indicated better results.
Time Frame: At Baseline and after 1 week, 4 weeks and 8 weeks
Population: Analysis was performed on mITT population which included all randomized participants who received at least one dose of study product and had at least one post randomization measure of gum comfort recorded via the questionnaire. Number analyzed included participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 59 | 58
Score on scale
  Change from baseline after week 1 | -0.5 (2.95) | -0.3 (1.67)
  Change from baseline after week 4: number analyzed (Participants) | 58 | 58
  Change from baseline after week 4 | -1.0 (3.46) | -0.2 (2.47)
  Change from baseline after week 8: number analyzed (Participants) | 58 | 58
  Change from baseline after week 8 | -1.0 (3.44) | -0.4 (3.34)

3. Secondary Outcome: Gum Health Analysis by Change From Baseline in Mean Scores of Participant Responses to the Individual Questions on the Gum Comfort Questionnaire After 1, 4, 8 and 12 Weeks.
Description: Gum comfort questionnaire was referred to assess the gum health of the denture wearer and to compare the ability of an experimental denture adhesive to provide self-perceived mucosal benefits compared to the use of no adhesive after 1, 4, 8 and 12 weeks of product use. It was comprised of 5 questions- Q1: My gums feel comfortable when wearing my denture(s), Q2: I feel my gums are cushioned from the impact of chewing and biting; Q3: My gums do not feel sore at the end of the day; Q4: My gums are not irritated by trapped food particles under my denture(s); Q5: My gums do not feel tired at the end of the day. The participants recorded the response on scale of 0-4: 0-Agree Strongly, 1-Agree Somewhat, 3-Neither Agree or Disagree, 4= Disagree Strongly). Total score range is 0-20 where lower score indicated better results.
Time Frame: At Baseline and after 1 week, 4 weeks, 8 weeks and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 59 | 58
Score on scale
  Q1: Baseline | 0.6 (0.95) | 0.6 (0.8)
  Q1: Change from BL after week 1 | -0.1 (0.86) | 0.1 (0.45)
  Q1: Change from BL after week 4: number analyzed (Participants) | 58 | 58
  Q1: Change from BL after week 4 | -0.1 (0.81) | 0.1 (0.66)
  Q1: Change from BL after week 8: number analyzed (Participants) | 58 | 58
  Q1: Change from BL after week 8 | -0.0 (0.84) | -0.1 (0.66)
  Q1: Change from BL after week 12: number analyzed (Participants) | 58 | 58
  Q1: Change from BL after week 12 | -0.1 (0.81) | 0.0 (0.95)
  Q2: Baseline | 0.9 (0.99) | 1.0 (0.79)
  Q2: Change from BL after week 1 | -0.1 (1.02) | -0.1 (0.76)
  Q2: Change from BL after week 4: number analyzed (Participants) | 58 | 58
  Q2: Change from BL after week 4 | -0.3 (1.05) | 0.1 (0.92)
  Q2: Change from BL after week 8: number analyzed (Participants) | 58 | 58
  Q2: Change from BL after week 8 | -0.1 (1.27) | 0.0 (1.23)
  Q2: Change from BL after week 12: number analyzed (Participants) | 58 | 58
  Q2: Change from BL after week 12 | -0.2 (1.20) | -0.0 (1.13)
  Q3: Baseline | 0.6 (0.99) | 0.6 (0.82)
  Q3: Change from BL after week 1 | 0.0 (0.78) | 0.1 (0.79)
  Q3: Change from BL after week 4: number analyzed (Participants) | 58 | 58
  Q3: Change from BL after week 4 | -0.1 (0.98) | 0.2 (0.85)
  Q3: Change from BL after week 8: number analyzed (Participants) | 58 | 58
  Q3: Change from BL after week 8 | -0.1 (0.88) | 0.2 (0.90)
  Q3: Change from BL after week 12: number analyzed (Participants) | 58 | 58
  Q3: Change from BL after week 12 | 0.0 (0.88) | 0.1 (1.11)
  Q4: Baseline | 1.3 (1.23) | 1.5 (1.05)
  Q4: Change from BL after week 1 | -0.2 (0.96) | -0.2 (0.88)
  Q4: Change from BL after week 4: number analyzed (Participants) | 58 | 58
  Q4: Change from BL after week 4 | -0.3 (1.01) | -0.4 (0.96)
  Q4: Change from BL after week 8: number analyzed (Participants) | 58 | 58
  Q4: Change from BL after week 8 | -0.4 (1.07) | -0.4 (1.08)
  Q4: Change from BL after week 12: number analyzed (Participants) | 58 | 58
  Q4: Change from BL after week 12 | -0.2 (1.01) | -0.3 (1.28)
  Q5: Baseline | 0.8 (1.05) | 0.8 (1.02)
  Q5: Change from BL after week 1 | -0.2 (1.05) | -0.1 (0.65)
  Q5: Change from BL after week 4: number analyzed (Participants) | 58 | 58
  Q5: Change from BL after week 4 | -0.2 (1.10) | -0.1 (0.77)
  Q5: Change from BL after week 8: number analyzed (Participants) | 58 | 58
  Q5: Change from BL after week 8 | -0.3 (1.03) | -0.1 (1.00)
  Q5: Change from BL after week 12: number analyzed (Participants) | 58 | 58
  Q5: Change from BL after week 12 | -0.2 (0.95) | -0.1 (1.12)

4. Secondary Outcome: Mucosal Health Analysis of Denture Bearing Tissues by Change From Baseline in Mucosal Score Assessment (MSA) After 1, 4, 8 and 12 Weeks
Description: MSA used by dentist to assess health of denture bearing tissues of participants across whole mouth on scale:1-4,1- normal appearance of gingiva,oral mucosa,2-mild inflammation(slight redness and/or hypertrophy/hyperplasia of gingiva and slight redness in some areas of palatal mucosa,including red spots indicating inflamed salivary duct orifices),3-moderate inflammation(marked redness and hypertrophy/hyperplasia of the gingiva, in large ares of palate, in oral mucosa, ulceration caused by denture, red and inflamed fibro-epithelial hyperplasia caused by denture),4-severe inflammation(severe redness and hypertrophy/hyperplasia of gingiva,spontaneous gingival bleeding, marked palatal granulations, inflamed oral mucosa areas).MSA was performed on denture-bearing tissues for either/both dentures across whole mouth and examiner recorded highest applicable score. Lower score indicated better results.
Time Frame: At Baseline and after 1 week, 4 weeks, 8 weeks and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 59 | 58
Score on scale
  Baseline | 1.8 (0.78) | 1.7 (0.71)
  Change from baseline after week 1 | -0.1 (0.55) | 0.0 (0.61)
  Change from baseline after week 4: number analyzed (Participants) | 58 | 58
  Change from baseline after week 4 | -0.2 (0.78) | -0.1 (0.66)
  Change from baseline after week 8: number analyzed (Participants) | 58 | 58
  Change from baseline after week 8 | -0.2 (0.73) | -0.1 (0.63)
  Change from baseline after week 12: number analyzed (Participants) | 58 | 58
  Change from baseline after week 12 | -0.3 (0.64) | -0.1 (0.65)

5. Secondary Outcome: Oral Health Related Quality of Life (OHrQoL) Analysis by Change From Baseline in Overall Mean Scores of Participant Responses to the Oral Health Impact Profile for Edentulous Patients (OHIP)-Edent Questionnaires After 1, 4, 8 and 12 Weeks
Description: OHIP-Edent questionnaire was used for the evaluation of OHrQoL. This questionnaire was comprised of 19 questions grouped into 6 functional domains and the participants responded on the scale of 0-4: 0-never, 1-rarely, 2-occasionally, 3-often and 4-very often. The functional domains are: domain 1- functional limitations (questions 1-3, score range 0-12), domain 2- physical pain (questions 4-7, score range 0-16), domain 3- psychological discomfort (questions 8-9, score range 0-8), domain 4- physical disability (questions 10-12, score range 0-12), domain 5- psychological disability (questions 13-14, score range 0-8) and domain 6- social disability (questions 15-19, score range 0-20). The overall score range is 0-76 where 0 is the best possible score. Lower scores represent a more favorable perception of participants OHrQoL.
Time Frame: At Baseline and after 1 week, 4 weeks, 8 weeks and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 59 | 58
Score on scale
  Baseline | 17.3 (12.79) | 15.7 (8.61)
  Change from baseline after week 1 | -2.7 (9.16) | -1.3 (3.72)
  Change from baseline after week 4: number analyzed (Participants) | 58 | 58
  Change from baseline after week 4 | -3.5 (9.32) | -1.9 (5.23)
  Change from baseline after week 8: number analyzed (Participants) | 58 | 58
  Change from baseline after week 8 | -3.6 (7.62) | -2.4 (5.85)
  Change from baseline after week 12: number analyzed (Participants) | 58 | 58
  Change from baseline after week 12 | -3.2 (8.23) | -2.9 (8.60)

6. Secondary Outcome: OHrQoL Analysis by Change From Baseline in Average Domain Scores of Participant Responses to the OHIP-Edent Questionnaires After 1, 4, 8 and 12 Weeks
Description: as for outcome 5
Time Frame: At Baseline and after 1 week, 4 weeks, 8 weeks and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 59 | 58
Score on scale
  Functional Limitations: Baseline (BL) | 3.6 (2.85) | 3.9 (2.01)
  Functional Limitations:Change from BL after week1 | -0.4 (2.25) | -0.6 (1.38)
  Functional Limitations:Change from BL after week4: number analyzed (Participants) | 58 | 58
  Functional Limitations:Change from BL after week4 | -0.7 (2.32) | -0.8 (1.75)
  Functional Limitations:Change from BL after week8: number analyzed (Participants) | 58 | 58
  Functional Limitations:Change from BL after week8 | -0.7 (2.04) | -0.9 (1.55)
  Functional Limitations:Change from BL after week12: number analyzed (Participants) | 58 | 58
  Functional Limitations:Change from BL after week12 | -0.7 (2.09) | -1.0 (2.09)
  Physical pain: Baseline | 3.6 (2.89) | 3.7 (2.43)
  Physical pain: Change from BL after week1 | -0.5 (2.31) | -0.3 (1.62)
  Physical pain: Change from BL after week4: number analyzed (Participants) | 58 | 58
  Physical pain: Change from BL after week4 | -0.8 (2.49) | -0.4 (1.75)
  Physical pain: Change from BL after week8: number analyzed (Participants) | 58 | 58
  Physical pain: Change from BL after week8 | -0.8 (2.07) | -0.4 (1.74)
  Physical pain: Change from BL after week12: number analyzed (Participants) | 58 | 58
  Physical pain: Change from BL after week12 | -0.7 (2.08) | -0.6 (2.50)
  Psychological (Psych) discomfort: Baseline | 2.1 (2.15) | 2.2 (1.74)
  Psych discomfort:Change from BL after week1 | -0.3 (1.85) | -0.4 (1.01)
  Psych discomfort:Change from BL after week4: number analyzed (Participants) | 58 | 58
  Psych discomfort:Change from BL after week4 | -0.2 (1.58) | -0.7 (1.22)
  Psych discomfort:Change from BL after week8: number analyzed (Participants) | 58 | 58
  Psych discomfort:Change from BL after week8 | -0.3 (1.62) | -0.7 (1.24)
  Psych discomfort:Change from BL after week12: number analyzed (Participants) | 58 | 58
  Psych discomfort:Change from BL after week12 | -0.2 (1.38) | -0.8 (1.56)
  Physical disability: Baseline | 3.2 (2.60) | 2.5 (1.91)
  Physical disability:Change from BL after week1 | -0.3 (2.14) | -0.1 (1.14)
  Physical disability:Change from BL after week4: number analyzed (Participants) | 58 | 58
  Physical disability:Change from BL after week4 | -0.5 (2.06) | -0.2 (1.39)
  Physical disability:Change from BL after week8: number analyzed (Participants) | 58 | 58
  Physical disability:Change from BL after week8 | -0.7 (1.74) | -0.3 (1.69)
  Physical disability:Change from BL after week12: number analyzed (Participants) | 58 | 58
  Physical disability:Change from BL after week12 | -0.7 (2.15) | -0.4 (1.90)
  Psychological (Psych) disability: Baseline | 1.8 (2.09) | 1.6 (1.33)
  Psych disability:Change from BL after week1 | -0.4 (1.65) | 0.0 (0.92)
  Psych disability:Change from BL after week4: number analyzed (Participants) | 58 | 58
  Psych disability:Change from BL after week4 | -0.4 (1.65) | -0.2 (1.05)
  Psych disability:Change from BL after week8: number analyzed (Participants) | 58 | 58
  Psych disability:Change from BL after week8 | -0.5 (1.48) | -0.3 (1.03)
  Psych disability:Change from BL after week12: number analyzed (Participants) | 58 | 58
  Psych disability:Change from BL after week12 | -0.4 (1.77) | -0.4 (1.27)
  Social disability: Baseline | 2.9 (3.17) | 1.9 (2.39)
  Social disability:Change from BL after week1 | -0.7 (2.37) | 0.1 (1.13)
  Social disability:Change from BL after week4: number analyzed (Participants) | 58 | 58
  Social disability:Change from BL after week4 | -0.9 (2.20) | 0.4 (1.97)
  Social disability:Change from BL after week8: number analyzed (Participants) | 58 | 58
  Social disability:Change from BL after week8 | -0.6 (2.09) | 0.2 (1.99)
  Social disability:Change from BL after week12: number analyzed (Participants) | 58 | 58
  Social disability:Change from BL after week12 | -0.4 (2.30) | 0.3 (2.32)

7. Secondary Outcome: OHrQoL Analysis by Change From Baseline in Overall Mean Scores of Participant Responses to the General Oral Health Assessment Index (GOHAI) Questionnaires After 1, 4, 8 and 12 Weeks
Description: GOHAI questionnaire was used for the evaluation of OHrQoL. It was comprised of 12 questions with 6 possible responses. The participants responded on the scale of 0-5: 0-always, 1-very often, 2-often, 3-sometimes, 4-seldom and 5-never. The functional domain of the questionnaire are as: domain 1: functional (questions 1-4, score range 0-20, participant's ability to eat, speak and swallow); domain 2: psychological (questions 6,7,9-11, score range 0-25, participant's concerns, relationships and appearance); domain 3- pain/ discomfort (questions 5,8,12, score range 0-15, participant's discomfort during chewing, sensitivity to hot/cold/sweets and use of medications to manage oral pain). The responses were scored on a 0 (always)-5 (never) scale for all questions except 3, 5 and 7 where the scoring is reversed, and thus the range of scores for the questionnaire is 0-60, where 60 is the best possible score. Higher score indicated better results.
Time Frame: At Baseline and after 1 week, 4 weeks, 8 weeks and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 59 | 58
Score on scale
  Baseline | 46.3 (8.16) | 48.6 (6.93)
  Change from baseline after week 1 | 0.8 (5.89) | 0.2 (3.57)
  Change from baseline after week 4: number analyzed (Participants) | 58 | 58
  Change from baseline after week 4 | 1.9 (6.34) | 0.7 (5.55)
  Change from baseline after week 8: number analyzed (Participants) | 58 | 58
  Change from baseline after week 8 | 2.9 (6.20) | 1.1 (6.19)
  Change from baseline after week 12: number analyzed (Participants) | 58 | 58
  Change from baseline after week 12 | 2.5 (7.38) | 0.9 (6.82)

8. Secondary Outcome: OHrQoL Analysis by Change From Baseline in Average Domain Scores of Participant Responses to the GOHAI Questionnaires After 1, 4, 8 and 12 Weeks
Description: as for outcome 7
Time Frame: At Baseline and after 1 week, 4 weeks, 8 weeks and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 59 | 58
Score on scale
  Functional domain: Baseline (BL) | 14.9 (3.63) | 15.8 (3.11)
  Functional domain:Change from BL after week1 | 0.6 (3.21) | -0.1 (1.92)
  Functional domain:Change from BL after week4: number analyzed (Participants) | 58 | 58
  Functional domain:Change from BL after week4 | 0.9 (3.07) | 0.7 (2.86)
  Functional domain:Change from BL after week8: number analyzed (Participants) | 58 | 58
  Functional domain:Change from BL after week8 | 1.2 (3.28) | 0.7 (2.95)
  Functional domain:Change from BL after week12: number analyzed (Participants) | 58 | 58
  Functional domain:Change from BL after week12 | 1.3 (2.99) | 0.8 (3.17)
  Psychosocial domain: Baseline | 20.1 (4.34) | 20.9 (3.44)
  Psychosocial domain:Change from BL after week1 | -0.2 (2.89) | 0.2 (1.56)
  Psychosocial domain:Change from BL after week4: number analyzed (Participants) | 58 | 58
  Psychosocial domain:Change from BL after week4 | 0.7 (3.97) | 0.1 (2.77)
  Psychosocial domain:Change from BL after week8: number analyzed (Participants) | 58 | 58
  Psychosocial domain:Change from BL after week8 | 1.1 (3.68) | 0.3 (2.98)
  Psychosocial domain:Change from BL after week12: number analyzed (Participants) | 58 | 58
  Psychosocial domain:Change from BL after week12 | 0.6 (3.89) | 0.3 (3.49)
  Pain/Discomfort domain: Baseline | 11.3 (2.49) | 11.8 (2.12)
  Pain/Discomfort domain:Change from BL after week1 | 0.4 (1.73) | 0.1 (2.03)
  Pain/Discomfort domain:Change from BL after week4: number analyzed (Participants) | 58 | 58
  Pain/Discomfort domain:Change from BL after week4 | 0.3 (2.52) | -0.0 (1.96)
  Pain/Discomfort domain:Change from BL after week8: number analyzed (Participants) | 58 | 58
  Pain/Discomfort domain:Change from BL after week8 | 0.7 (2.27) | 0.1 (2.16)
  Pain/Discomfort domain:Change from BL after week12: number analyzed (Participants) | 58 | 58
  Pain/Discomfort domain:Change from BL after week12 | 0.6 (2.90) | -0.3 (2.42)

9. Secondary Outcome: Mean Scores of Participant Responses to the Sensory Questionnaire at Week 4
Description: Sensory attributes of the adhesive was assessed by sensory questionnaire which was comprised of 6 questions; Q1: I feel the product has a smooth texture on my gums, Q2: I feel the product is gentle on my gums, Q3: I feel the product flavor soothes my gums, Q4: I feel the product flavor cools my gums, Q5: I feel the product is easy to apply, Q6: I feel less rubbing from my denture throughout the day when using this product. This questionnaire was only referred to participants randomized to the experimental adhesive group. The participants responded for all questions on the scale of 0-4: 0-agree strongly,1-agree somewhat, 2-neither agree or disagree, 3-disagree somewhat, 4-disagree strongly. The total score range is 0-24 where a low score indicated better results.
Time Frame: At week 4
Population: Analysis was performed on mITT population of only experimental denture adhesive group. Number analyzed included participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 59 | 0
Score on scale | 4.7 (3.30) |

ADVERSE EVENTS:
Time Frame: From signing of the informed consent form until 5 days after last administration of study drug (or last procedure).
Description: Safety population included all participants who were randomized and received at least one dose of investigational product. All adverse events (AEs) were summarized by system organ class and preferred term. All treatment emergent AEs and serious AEs were collected and reported.
Groups:
- Overall: Included all participants that were assessed for safety adverse events.
Arm/Group | Experimental Denture Adhesive | No Adhesive | Overall
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59 | 0/119
Other Adverse Events (participants affected / at risk) | 30/60 | 19/59 | 49/119
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Denture Adhesive (N=60) | No Adhesive (N=59) | Overall (N=119)
Oral mucosal erythema (Gastrointestinal disorders) | 14 (16) | 15 (16) | 29 (32)
Gingival erythema (Gastrointestinal disorders) | 14 (14) | 7 (8) | 21 (22)
Salivary duct inflammation (Gastrointestinal disorders) | 3 (3) | 5 (5) | 8 (8)
Oral mucosal hypertrophy (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gingival ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Palatal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03807700/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03807700/SAP_001.pdf